CLINICAL TRIAL: NCT02443298
Title: Phase IIa, Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Assess the Safety and Efficacy of Subcutaneously Administered BI 655066/ABBV-066 (Risankizumab) as add-on Therapy Over 24 Weeks in Patients With Severe Persistent Asthma.
Brief Title: Efficacy and Safety of BI 655066/ABBV-066 (Risankizumab) in Patients With Severe Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1311.14; 2014-004932-20 (EudraCT Number)
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Risankizumab (Experimental): Patients received subcutaneous injection of 1 milliliter (mL) prefilled syringe with 90 milligram/ milliliter (mg/mL) risankizumab once every 4 weeks (weeks 0, 4, 8, 12, 16, 20).
  Interventions: Drug: risankizumab
- Placebo (Placebo Comparator): Patients received subcutaneous injection of 1 milliliter (mL) prefilled syringe consisting of matching placebo to risankizumab once every 4 weeks (weeks 0, 4, 8, 12, 16, 20).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Matching placebo for risankizumab
  Arms: Placebo
Drug: risankizumab — Monoclonal IgG antibody
  Other Names: ABBV-066; BI 655066
  Arms: Risankizumab

SUMMARY:
The objectives of this trial are primarily to evaluate the efficacy and safety of BI 655066/ABBV-066 (risankizumab) as compared to placebo over a 24-week treatment period in severe asthma patients. The primary endpoint is time to first asthma worsening during the planned 24 week treatment period for active vs. placebo treated patients on top of standard of care therapy. Upon demonstration of a meaningful clinical response, another important objective is the identification of biomarkers that can be used to target patients who will likely respond to treatment with BI 655066/ABBV-066 (risankizumab).

ELIGIBILITY:
Inclusion criteria:

1. Pre-bronchodilator clinic measured forced expiratory volume (FEV1) of =40% and =85% of predicted normal.
2. One year history of asthma diagnosed by a physician, and have FEV1 reversibility of =12% and an absolute change of at least 200 mL after administration of 400 µg salbutamol.
3. Must be on at least medium dose inhaled corticosteroids and at least one other asthma controller medication for at least one year.
4. Must have documented history of two or more severe asthma exacerbations in the last 12 months.

Exclusion criteria:

1. Patients with a significant disease other than asthma.
2. Patients who are not able to produce sputum or sputum samples of sufficient quality.
3. Patients who had clinically relevant history of intubation for asthma exacerbation in the past year.
4. Patients diagnosed with any concurrent respiratory disease.
5. Recent history (within 6 months) of myocardial infarction or hospitalized for cardiac failure in the past year.
6. Patients who have undergone thoracotomy with pulmonary resection.
7. Patients who have undergone bronchial thermoplasty or radiotherapy procedure in the past year or have planned procedures during the study.
8. Patients taking oral corticosteroids with a total daily dose of more than 20 mg prednisone (or equivalent) in the past 6 weeks.
9. Pregnant or nursing women.
10. Women of childbearing potential that, if sexually active, is unwilling to use a highly effective method of birth control.
11. Clinically relevant acute infections or chronic infections.
12. Have received any live bacterial or live viral vaccination in the last12 weeks.
13. Have received Bacille Calmette-Guerin (BCG) vaccination in the last 12 months.
14. Have received treatment with ustekinumab (Stelara®).
15. Have received treatment with any other biologics in the last 3 months or within 6 times the half-life of the compound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (64):
- United States (20):
  - WCCT Global, LLC, Costa Mesa, California
  - El Camino Hospital, Mountain View, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - VA WNY Healthcare System, Buffalo, New York
  - American Health Research, Inc., Charlotte, North Carolina
  - Coastal Carolina Health Care, P.A., New Bern, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Research Protocol Mgmt Spc, Pittsburgh, Pennsylvania
  - MedTrial, LLC, Columbia, South Carolina
  - VitaLink Research, Greenville, South Carolina
  - Respiratory and Sleep Disorders Specialists, The Woodlands, Texas
  - O and O Alpan, LLC, Fairfax, Virginia
- Belgium (4):
  - ULB Hopital Erasme, Brussels
  - Brussels - UNIV St-Luc, Brussels
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Burlington Lung Clinic, Burlington, Ontario
  - Airway Inflammometry Laboratory, Hamilton, Ontario
- France (5):
  - HOP CHU de Grenoble, Grenoble
  - HOP Nord, Marseille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Nord Laënnec, Nantes
  - HOP Bichat, Paris
- Germany (15):
  - Praxis Dr. Linnhoff, Berlin, Berlin
  - MECS Research GmbH, Berlin, Berlin
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil gGmbH, Bochum
  - Praxis Dr. med. Claus Keller, Frankfurt
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Medaimun GmbH, Frankfurt
  - Hamburger Institut für Therapieforschung GmbH (HIT), Hamburg
  - Praxis Dr. Hoffmann, Hannover, Hanover
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - KPPK GmbH, Studienzentrum, Koblenz
  - KLB Gesundheitsforschung Lübeck GmbH, Lübeck
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Institut für klinische Forschung GmbH, Neu-Isenburg
  - IFG Institut für Gesundheitsförderung GmbH, Rüdersdorf
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - HagaZiekenhuis, The Hague
- Poland (4):
  - Gibinski Univ.Clin.Cnter of Silesian Med.Uni.Katowice,Outpat, Katowice
  - Specjalistyczny Osrodek Alergologiczno-Intern. ALL-MED, Krakow
  - Univ. Hospital in Krakow,Pulmonology Clinical Dept, Krakow
  - Barlicki University Hospital No. 1, Lodz
- South Korea (4):
  - Chungbuk National University Hospital, Cheongju-si
  - Chonnam National University Hospital, Gwangju
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, St.Paul's Hospital, Seoul
- Taiwan (2):
  - Chang Gung Memorial Hospital Keelung, Keelung
  - China Medical University Hospital, Taichung
- United Kingdom (5):
  - Celerion Inc, Belfast
  - Bradford Royal Infirmary, Bradford
  - Glenfield Hospital, Leicester
  - The Medicines Evaluation Unit, Manchester
  - Wishaw General Hospital, Wishaw

REFERENCES:
- [Derived] Brightling CE, Nair P, Cousins DJ, Louis R, Singh D. Risankizumab in Severe Asthma - A Phase 2a, Placebo-Controlled Trial. N Engl J Med. 2021 Oct 28;385(18):1669-1679. doi: 10.1056/NEJMoa2030880. PMID 34706172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, parallel-group multicenter study to assess the efficacy and safety of risankizumab, an IL-23p19 monoclonal antibody, compared to placebo in patients with severe persistent asthma.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended a specialist sites which ensured that they (the patients) met all strictly implemented inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any one of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | Risankizumab | Placebo
Started | 105 | 109
Completed | 101 | 104
Not Completed | 4 | 5
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Set (RS): This patient set included all randomized patients, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risankizumab | Placebo | Total
Number analyzed (Participants) | 105 | 109 | 214
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (11.3) | 52.3 (12.5) | 53.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 64 | 133
  Male | 36 | 45 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 102 | 106 | 208
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 11 | 11 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 84 | 88 | 172
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Oral corticosteroid (OCS) use at baseline [Count of Participants; unit: Participants]
  Yes | 15 | 17 | 32
  No | 90 | 92 | 182
Baseline Morning peak expiratory flow (PEF) [Mean (Standard Deviation); unit: Liter/Minute (L/min)] | 299.34 (110.50) | 309.56 (115.34) | 304.54 (112.84)
Baseline 24 Hour Rescue Medication Use [Mean (Standard Deviation); unit: Puff] — Baseline 24 Hour Rescue Medication Use: Average over the 14 days prior to randomization
  Puff | 3.17 (3.81) | 3.89 (4.78) | 3.53 (4.34)
Baseline First 5 questions of the Asthma Control Questionnaire (ACQ5) Score [Mean (Standard Deviation); unit: Unit on scale] — Baseline ACQ5 is the mean of last 2 available measurements in last 2 weeks prior to Visit 2, that is, 14 days prior to the administration of the first dose. Weekly score is average of responses to the five questions. ACQ5 asks patients to rate the severity of their asthma symptoms and the degree to which asthma affected their sleep and other daily activities. The scale for all five questions range from the best possible answer of 0 (No symptoms, None, Never) to the worst possible answer of 6 (very severe, unable to sleep, totally limited). ACQ5 score can range from 0.0 (best) to 6.0 (worst).
  Unit on scale | 2.15 (1.15) | 2.39 (1.17) | 2.27 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Asthma Worsening During the Planned 24 Week Treatment Period
Description: Time to first asthma worsening during the planned 24 week treatment period:
  Asthma worsening was defined as the occurrence of any one of the following four criteria:
  a) Decrease from baseline of ≥30% in morning peak expiratory flow (PEF) on at least 2 consecutive days. b) Increase from baseline of ≥50% and an increase of least 4 puffs in daily use of rescue medication for at least 2 consecutive days. c) Increase from baseline of ≥0.75 units in ACQ5. d) Severe asthma exacerbations defined as initiation of systemic corticosteroids (prednisone or equivalent) for 3 or more consecutive days for asthma. Additionally, for subjects on maintenance systemic corticosteroids, at least doubling of the maintenance dose resulting in a total daily dose of ≥ 20 mg for three or more consecutive days was considered a severe asthma exacerbation.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of treatment.
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Days | 40.00 [30.00 to 52.00] | 85.50 [63.00 to 131.00]
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; This was analyzed by using a Cox proportional hazards model that included treatment and the stratification factor of OCS use at baseline as fixed effects; Test type: Superiority; p = 0.0255, Cox proportional hazards model; Hazard Ratio (HR) = 1.46, 80% CI 2-sided [1.18 to 1.81] — Comparison of Risankizumab to Placebo

2. Secondary Outcome: Time to First Asthma Worsening During the Planned 24 Week Treatment Period According to Alternative Definition
Description: Time to first asthma worsening during the planned 24 week treatment period according to alternative definition:
  Asthma worsening was defined as the occurrence of any one of the following four criteria:
  a) Decrease from baseline of ≥30% in morning peak expiratory flow (PEF) on at least 2 consecutive days. b) Increase from baseline of ≥50% and an increase of least 4 puffs in daily use of rescue medication for at least 2 consecutive days. c) Increase from baseline of ≥0.5 units in ACQ5. d) Severe asthma exacerbations defined as initiation of systemic corticosteroids (prednisone or equivalent) for 3 or more consecutive days for asthma. Additionally, for subjects on maintenance systemic corticosteroids, at least doubling of the maintenance dose resulting in a total daily dose of ≥ 20 mg for three or more consecutive days was considered a severe asthma exacerbation.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of treatment.
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Days | 20.00 [16.00 to 25.00] | 37.00 [31.00 to 45.00]
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0131, Cox proportional hazards model; Hazard Ratio (HR) = 1.47, 80% CI 2-sided [1.20 to 1.79] — Comparison of Risankizumab to Placebo

3. Secondary Outcome: Annualized Rate of Asthma Worsening During the Planned 24 Week Treatment Period
Description: Annualized rate of asthma worsening during the planned 24 week treatment period.
  Asthma worsening was defined as the occurrence of any one of the following four criteria:
  a) Decrease from baseline of ≥30% in morning peak expiratory flow (PEF) on at least 2 consecutive days. b) Increase from baseline of ≥50% and an increase of least 4 puffs in daily use of rescue medication for at least 2 consecutive days. c) Increase from baseline of ≥0.75 units in ACQ5. d) Severe asthma exacerbations defined as initiation of systemic corticosteroids (prednisone or equivalent) for 3 or more consecutive days for asthma. Additionally, for subjects on maintenance systemic corticosteroids, at least doubling of the maintenance dose resulting in a total daily dose of ≥ 20 mg for three or more consecutive days was considered a severe asthma exacerbation.
  Mean is Annualized rate.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of treatment.
Measure: Mean (Standard Error); unit: Events per patient year
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Events per patient year | 4.8412 (0.577) | 3.2410 (0.401)
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; Annualized rate is obtained from fitting a negative binomial regression including logarithm of the exposure as an offset, treatment, and OCS use at baseline as covariate; Test type: Superiority; p = 0.0065, Negative binomial regression; Rate Ratio = 1.4937, 80% CI 2-sided [1.2366 to 1.8044], Standard Error of Mean 0.220 — Comparison of Risankizumab to Placebo

4. Secondary Outcome: Time to First Severe Asthma Exacerbation During the Planned 24 Week Treatment Period
Description: Time to first severe asthma exacerbation during the planned 24 week treatment period. Severe asthma exacerbation was defined as initiation of systemic corticosteroids (prednisone or equivalent) for 3 or more consecutive days for asthma. Additionally, for subjects on maintenance systemic corticosteroids, at least doubling of the maintenance dose resulting in a total daily dose of ≥ 20 mg for three or more consecutive days was considered a severe asthma exacerbation.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of treatment. NA = not estimable due to an insufficient numbers of patient with an event
Measure: Median (80% Confidence Interval); unit: Days
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Days | NA [NA to NA] — Not estimable due to an insufficient numbers of patient with an event | NA [NA to NA] — Not estimable due to an insufficient numbers of patient with an event
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; Time to first event is obtained from fitting a Cox proportional-hazards model including treatment, and OCS use at baseline as covariate; Test type: Superiority; p = 0.4619, Cox proportional hazards model; Hazard Ratio (HR) = 1.18, 80% CI 2-sided [0.88 to 1.57] — Comparison of Risankizumab to Placebo

5. Secondary Outcome: Annualized Rate of Severe Asthma Exacerbation During the Planned 24-week Treatment Period
Description: Annualized rate of severe asthma exacerbation during the planned 24-week treatment period.
  Severe asthma exacerbation was defined as initiation of systemic corticosteroids (prednisone or equivalent) for 3 or more consecutive days for asthma. Additionally, for subjects on maintenance systemic corticosteroids, at least doubling of the maintenance dose resulting in a total daily dose of ≥ 20 mg for three or more consecutive days was considered a severe asthma exacerbation.
  Mean is Annualized rate.
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of treatment.
Measure: Mean (Standard Error); unit: Events per patient year
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Events per patient year | 1.5901 (0.257) | 1.4051 (0.228)
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.5550, Negative binomial regression; Rate Ratio = 1.1317, 80% CI 2-sided [0.8652 to 1.4803], Standard Error of Mean 0.237 — Comparison of Risankizumab to Placebo

6. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) In-clinic Change From Baseline at Week 24
Description: Trough forced expiratory volume in 1 second (FEV1) in-clinic change from baseline at week 24.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of treatment. One patient not included in the analysis due to missing baseline value. Number of patients with either baseline or on-treatment data at the respective week and does not require having both.
Measure: Least Squares Mean (Standard Error); unit: Liter (L)
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Liter (L) | -0.052 (0.036) | -0.013 (0.035)
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; The adjusted mean (SE) are obtained from fitting a mixed effect repeated measures (MMRM) model including treatment, OCS use at baseline, test day, treatment-by-test day interaction, baseline, and baseline-by-test day interaction as covariates patient as a random effect; Test type: Superiority; p = 0.4423, Mixed Models Analysis; Unstructured covariance structure for within-patient variation; Mean Difference (Final Values) = -0.039, 80% CI 2-sided [-0.104 to 0.026], Standard Error of Mean 0.051 — Comparison of Risankizumab to Placebo

7. Secondary Outcome: Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) In-clinic Change From Baseline at Week 24
Description: Post-bronchodilator forced expiratory volume in 1 second (FEV1) in-clinic change from baseline at week 24.
Time Frame: Baseline and 24 weeks
Population: FAS: All randomized patients who received at least one dose of treatment. One patient not included in the analysis due to missing baseline value and one patient not included in the analysis due to missing on-treatment data. Number of patients with either baseline or on-treatment data at the respective week and does not require having both.
Measure: Least Squares Mean (Standard Error); unit: Liter (L)
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Liter (L) | -0.097 (0.032) | -0.030 (0.032)
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.1377, Mixed Models Analysis; Unstructured covariance structure for within-patient variation; Mean Difference (Final Values) = -0.068, 80% CI 2-sided [-0.126 to -0.009], Standard Error of Mean 0.045 — Comparison of Risankizumab to Placebo

8. Secondary Outcome: Weekly Asthma Control Questionaire Score at Week 24
Description: The score at week 24 is the average of the responses to the five ACQ5 questions for the week preceding the Week 24 visit. The ACQ5 asks patients to rate the severity of their asthma symptoms and the degree to which asthma affected their sleep and other daily activities. The scale for all five ACQ5 questions range from the best possible answer of 0 (No symptoms, None, Never) to the worst possible answer of 6 (very severe, unable to sleep, totally limited). The ACQ5 score can range from 0.0 (best) to 6.0 (worst).
Time Frame: 24 weeks
Population: Full Analysis Set (FAS): All randomized patients who received at least one dose of treatment. Ten patients excluded from the analysis due to missing data at week 24.
Measure: Least Squares Mean (Standard Error); unit: Unit on Scale
Arm/Group | Risankizumab | Placebo
Number analyzed (Participants) | 105 | 109
Unit on Scale | 1.857 (0.099) | 1.708 (0.099)
Statistical Analysis 1: Comparison: Risankizumab vs Placebo; The adjusted mean (SE) are obtained from fitting an analysis of covariance (ANCOVA) model separately for each week including treatment, OCS use at baseline, and baseline as covariates. The weekly averages of daily measurements are calculated before fitting the model; Test type: Superiority; p = 0.1985, ANCOVA; Mean Difference (Final Values) = 0.149, 80% CI 2-sided [0.000 to 0.297], Standard Error of Mean 0.115 — Comparison of Risankizumab to Placebo

ADVERSE EVENTS:
Time Frame: From the administration of first dose of study medication until 16 weeks after last dose of study medication, up to 40 weeks.
Arm/Group | Risankizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/109
Serious Adverse Events (participants affected / at risk) | 14/105 | 21/109
Other Adverse Events (participants affected / at risk) | 84/105 | 80/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risankizumab (N=105) | Placebo (N=109)
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risankizumab (N=105) | Placebo (N=109)
Bronchitis (Infections and infestations) | 11 | 9
Nasopharyngitis (Infections and infestations) | 11 | 22
Sinusitis (Infections and infestations) | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 9 | 10
Urinary tract infection (Infections and infestations) | 5 | 6
Blood creatine phosphokinase increased (Investigations) | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 6
Headache (Nervous system disorders) | 7 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 65 | 58
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT02443298/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02443298/SAP_001.pdf